CLINICAL TRIAL: NCT01888848
Title: Effects of Dietary Blueberry Supplementation on Cognition and Mobility in Healthy Older Adults
Brief Title: Effects of Blueberry on Cognition and Mobility in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Human Nutrition Research Center on Aging (U.S. Federal Agency)
Collaborators: U.S. Highbush Blueberry Council (Other); Tufts University (Other)
Responsible Party: Principal Investigator, Barbara Shukitt-Hale, Research Psychologist, USDA Human Nutrition Research Center on Aging
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USDAHNRC-2013-1; 1950-51000-070-19R (Other Grant/Funding Number: USHBC)
Record Dates: First submitted 2013-06-13; First posted 2013-06-28 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Aging; Age-Related Memory Disorders
Keywords: Postural Balance; Walking; Gait; Cognition; Learning; Memory; Blueberry; Antioxidants; Anti-Inflammatory Agents; Brain
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- blueberry (Experimental): Participants randomized into this arm of the study consume freeze-dried blueberry.
  Interventions: Dietary Supplement: Freeze-dried Blueberry
- placebo (Placebo Comparator): Participants randomized into this arm of the study consume a blueberry placebo.
  Interventions: Dietary Supplement: Blueberry Placebo

INTERVENTIONS:
Dietary Supplement: Freeze-dried Blueberry — 12g freeze-dried blueberry (powder), twice daily with water, for 90 days
  Arms: blueberry
Dietary Supplement: Blueberry Placebo — 12g blue, blueberry-flavored powder, twice daily with water, for 90 days
  Arms: placebo

SUMMARY:
This study is being conducted to assess the effect of dietary blueberry supplementation on cognition and mobility in older adults. It is hypothesized that plant compounds, present in blueberries, may improve cognition and mobility by protecting against oxidative stress and inflammation.

DETAILED DESCRIPTION:
This study is being conducted to assess the effect of dietary blueberry supplementation vs. placebo on measures of cognition and mobility in older adults. Participants will visit the HNRCA on 4 occasions. During the first visit, participants will complete a dietary assessment and familiarize themselves with some of the cognitive tests used in the study. After a period of up to 45 days participants will return for the second visit. Participants will be randomized to consume either freeze dried blueberry powder or a placebo powder that tastes like blueberry. At visits 2, 3 and 4, participants will undergo tests of cognition, memory, gait and balance. In addition, blood samples and 24-hour urine will be collected at these visits. Tests include balance and gait assessment using a treadmill instrumented with pressure sensors which will measure postural sway and a variety of spatial/temporal gait parameters. Participants will also be affixed with surface electrodes to measure the activation of muscles in their legs during these balance and gait measurements. Participants will complete a battery of cognitive tests on paper and by computer. In the time between participants' visit 2 and visit 4, participants will receive a weekly telephone call to check in with them and remind them to continue taking the study powder. At the very end of the study, when all participants are finished, participants will receive a telephone call to debrief them and notify them which group they were randomized into. An optional tissue banking protocol will be offered for collection of additional blood to be banked at visits 2-4.

ELIGIBILITY:
Inclusion Criteria:

* Men and women are between the ages of 60 and 75 years
* Body mass index 18.5-29.9 kg/m2
* Adequate visual acuity or corrected visual acuity to read and perform computer tasks.
* Fluency in spoken and written English
* Ability to walk independently for 20 minutes
* Absence of menstruation for a minimum of 12 months or surgical menopause.

Exclusion Criteria:

* Self-reported vegetarian or vegan.
* Any condition that has resulted in cognitive deficits, including but not limited to Alzheimer's disease or other dementias, cerebrovascular accident, or head injury
* History of any neurologic disorder resulting in permanent or relapsing/remitting neurologic impairment including but not limited to Parkinson's disease, amyotrophic lateral sclerosis, Huntington's disease, peripheral neuropathy, or radiculopathy.
* History of any condition resulting in permanent muscle or mobility deficit that would interfere with walking independent of assistance for 20 minutes, including but not limited to amputation, fracture, arthritis, myopathy, or limb, hip or back surgery within the last year.
* Self-reported cognitive, memory, neurologic or functional deficits that are stated to interfere with activities of daily living or functional status.
* Any chronic condition associated with increased risk of falls such as vestibular disease, orthostatic hypotension or neuropathy.
* Falls within the last year, that occurred in the course or routine daily activities, which were not precipitated by unusual circumstances such as being pushed or falling on ice.
* Regular use (i.e. that cannot or should not be discontinued for the entire study period, as per the subject's personal physician) of medications or dietary supplements known or suspected to influence cognitive function, attention, ability to ambulate, gait, balance, or risk of falls that in the opinion of the study physician may influence study results or increase risk with participation in the study.
* Psychiatric disorders that could in the opinion of the study physician interfere with study testing, including bipolar disorder, psychosis, and major depression
* MMSE score of less than 24 at screening
* Gastrointestinal disorders that influence digestion and absorption of food
* Diabetes mellitus
* Liver dysfunction
* History of cirrhosis
* SGPT, SGOT, or total bilirubin > 2 x upper limit of normal
* Kidney disease as indicated by serum creatinine > 1.5 mg/dL at screening
* Cardiac or pulmonary conditions that limit ambulation or results in dyspnea with ambulation with walking required as part of activities of daily living.
* Reported allergy to blueberry or ingredients in the placebo.
* Ethanol use estimated to be on average > 2 servings/day of beer (12-ounces), wine (5 ounces) or liquor (1.5 ounces), or self-reported binge-drinking.
* Illicit drug use in the last 12 months.
* Cigarette smoking within the last 6 months or current use of nicotine.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
cognition | change from baseline at 45 days
  Spatial memory and learning (Morris water maze); short-term memory (digit span), verbal learning and memory (California verbal learning Test), executive function (trail making test, task switching test), attention (attention network test)
cognition | Change from baseline at 90 days
  Spatial memory and learning (Morris water maze); short-term memory (digit span), verbal learning and memory (California verbal learning Test), executive function (trail making test, task switching test), attention (attention network test)

SECONDARY OUTCOMES:
Gait | Change from baseline at 90 days
  gait speed, step length variability, step width variability via instrumented treadmill
Gait | Change from baseline at 45 days
  gait speed, step length variability, step width variability via instrumented treadmill

OTHER OUTCOMES:
Balance | Change from baseline at 45 days
  sway velocity and sway area via pressure-sensor
Balance | Change from baseline at 90 days
  sway velocity and sway area via pressure-sensor

CONTACTS AND LOCATIONS:
Overall Officials: Edward Saltzman, MD, Principal Investigator — Tufts University; Barbara Shukitt-Hale, PhD, Study Director — United States Department of Agriculture (USDA)
Locations (1):
- Jean Meyer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Miller MG, Shukitt-Hale B. Berry fruit enhances beneficial signaling in the brain. J Agric Food Chem. 2012 Jun 13;60(23):5709-15. doi: 10.1021/jf2036033. Epub 2012 Feb 3. PMID 22264107
- [Background] Joseph JA, Shukitt-Hale B, Denisova NA, Bielinski D, Martin A, McEwen JJ, Bickford PC. Reversals of age-related declines in neuronal signal transduction, cognitive, and motor behavioral deficits with blueberry, spinach, or strawberry dietary supplementation. J Neurosci. 1999 Sep 15;19(18):8114-21. doi: 10.1523/JNEUROSCI.19-18-08114.1999. PMID 10479711
- [Background] Krikorian R, Shidler MD, Nash TA, Kalt W, Vinqvist-Tymchuk MR, Shukitt-Hale B, Joseph JA. Blueberry supplementation improves memory in older adults. J Agric Food Chem. 2010 Apr 14;58(7):3996-4000. doi: 10.1021/jf9029332. PMID 20047325
- See also: Human Nutrition Research Center on Aging at Tufts University website — http://hnrca.tufts.edu/
- See also: USDA ARS website — http://www.ars.usda.gov/main/main.htm
- See also: US Highbush Blueberry Council website — http://www.blueberry.org/